CLINICAL TRIAL: NCT02269475
Title: A Phase 3 Randomized, Double-blind Study to Evaluate the Efficacy and Safety of MEDI3250 Compared to Placebo in Healthy Japanese Children Age 7 Years Through 18 Years
Brief Title: A Phase3 Study to Evaluate the Efficacy and Safety of MEDI3250 in Healthy Japanese Children Age 7 Years Through 18 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: D2560C00006
Record Dates: First submitted 2014-10-13; First posted 2014-10-21 (Estimated); Results first posted 2015-12-03 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-02

CONDITIONS: Healthy Japanese Children Age 7 Years Through 18 Years
Keywords: Efficacy; Safety; Tolerability; MEDI3250; Japanese children

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MEDI3250 (Experimental): MEDI3250 Nasal Spray
  Interventions: Drug: MEDI3250
- Placebo (Placebo Comparator): Placebo Nasal spray
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MEDI3250 — MEDI3250
  Arms: MEDI3250
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The study is designed to gather the efficacy, safety and tolerability data in Japanese children 7 to 18 years of age that would support approval of MEDI3250 in Japan.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo controlled, multicenter study will enrol 1008 subjects. The study is designed to gather the efficacy, safety and tolerability data in Japanese children 7 through 18 years of age that would support approval of MEDI3250 in Japan.

For children age 7 years through 18 years, the recommended dosage schedule for intranasal administration is 0.2 mL (0.1 mL per nostril). For children age 7 years through 8 years not previously vaccinated against seasonal influenza, a second dose should be given after an interval of at least 4 weeks.

For the efficacy endpoint, data will be gathered on the incidence of laboratory-confirmed influenza-like illness in the two treatment arms. Laboratory-confirmed influenza-like illness would include cases of influenza diagnosed using culture-confirmation and/or PCR-based methods.

For the safety and tolerability endpoint, data will be gathered on solicited symptoms, AEs and SAEs.

Subject will be randomized 2:1 to receive MEDI3250 or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Age 7 through 18 years of age at the time of randomization.
2. A written informed consent should be obtained from the subject's legally acceptable representative, and a written informed assent should be obtained from the subject if possible.
3. Available for illness visits at clinic during the influenza surveillance period.
4. Ability of the legal representative to understand and comply with the requirements of the protocol．
5. Parent/guardian available by telephone, email or etc．
6. Females of childbearing potential, unless surgically sterile (ie, bilateral tubal ligation, bilateral oophorectomy, or hysterectomy), has sterile male partner, is premenarchal, or practices abstinence, must have used an effective method of avoiding pregnancy (including oral, transdermal, or implanted contraceptives, intrauterine device, female condom with spermicide, diaphragm with spermicide, cervical cap with spermicide, or use of a condom with spermicide by the sexual partner) for 30 days prior to the first dose of investigational product, and must agree to continue using such precautions for 60 days after the final dose of investigational product.
7. A subject who is considered by the investigator to be at risk of pregnancy must also have a negative urine pregnancy test at screening and, if screening and Day 0 do not occur on the same day, on the day of vaccination prior to randomization. Investigator judgment is required to assess each subject's need for pregnancy testing.
8. Healthy by medical history and physical examination OR presence of stable underlying chronic medical condition for which hospitalization has not been required in the previous year.

Exclusion Criteria:

1. Subjects who were previously administered influenza vaccine in 2014-2015 influenza season
2. Previous randomisation in the present study
3. Participation in another clinical study with an investigational product during the last 3 month
4. Acute illness or evidence of significant active infection at randomization;
5. Fever ≥99.5°F (37.5°C) at randomization;
6. Any drug therapy from 15 days prior to randomization or expected drug therapy through 28 days post last dose with the exception of the following classes/types of medications, which are allowed:

   Contraceptives (change in contraceptive type or method is acceptable as long as guidelines are followed for prevention of pregnancy during change); Topical corticosteroids, calcineurin inhibitors, or antifungals for uncomplicated dermatitis; Chronic medications (including those taken on an as-needed basis) that have been well tolerated and were not initiated and/or did not have a dosage change within 90 days prior to randomization.
7. Current or expected receipt of immunosuppressive medications within a 28-day window around any dose, including an immunosuppressive dose of corticosteroids, which is defined as ≥20 mg/day of prednisone or its equivalent, given daily or on alternate days for ≥15 days (intranasal, intra-articular, and topical corticosteroids are permitted); Note: topical corticosteroids for uncomplicated dermatitis may be used throughout the study according to the judgment of the investigator; topical calcineurin inhibitors may be used in accordance with their package insert at entry and during study participation.
8. Any known immunosuppressive condition or immune deficiency disease including known or suspected infection with human immunodeficiency virus (HIV);
9. History of allergic disease or reactions likely to be exacerbated by any component of the investigational product including allergy to eggs, egg proteins, gentamicin, or gelatin or serious, life threatening, or severe reactions to previous influenza vaccinations;
10. Use of aspirin or salicylate-containing medications within 28 days prior to randomization or expected receipt through the entire study;
11. History of Guillain-Barré syndrome;
12. Use of antiviral agents with activity against influenza virus (including amantadine, rimantadine, oseltamivir, and zanamivir) within 28 days prior to first dose of investigational product or anticipated use of such agents in the study period;
13. Administration of any live virus vaccine within 30 days prior to enrolment, or if receipt of another live virus vaccine is expected within 30 days of any study vaccination;
14. Administration of any inactivated vaccine within 14 days prior to enrolment or if receipt of another inactivated vaccine is expected within 14 days of any study vaccination;
15. Receipt of any blood product within 90 days prior to vaccination or expected receipt during this study;
16. Pregnant or lactating female
17. Involvement in the planning and conduct of the study (applies to all AstraZeneca staff and staff at the study site as a legal representative)
18. Any condition that, in the opinion of the investigator, might interfere with the interpretation or evaluation of the vaccines.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1369 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masaki Yokohama, MD, Principal Investigator — Yokohama clinic; Toshiko Yamaguchi, MD, Principal Investigator — Yamaguchi Clinic; Haruo Maeta, MD, Principal Investigator — Maeta Pediatrics Clinic; Hideki Nakazawa, MD, Principal Investigator — HIGASHIKATSUYAMA nakazawa Naika allergy Internal Medicine; Atsushi Shibasaki, MD, Principal Investigator — Shibasaki internal medicine & Pediatrics Clinic; Yutaka Igarashi, MD, Principal Investigator — Igarashi Children's Clinic; Keiko Mitamura, MD, Principal Investigator — Eiju General Hospital; Satoshi Yamada, MD, Principal Investigator — Kyouai Clinic; Kiyoshi Niwa, MD, Principal Investigator — Niwa Family Clinic; Ryuta Ono, MD, Principal Investigator — Kanagawa HImawari Clinic; Eiji Kato, MD, Principal Investigator — Fukuiken Saiseikai Hospital; Toshikazu Takahashi, MD, Principal Investigator — Takahashi Clinic; Ryouta Yoshimura, MD, Principal Investigator — Yoshimura Children's Clinic; Hiroshi Taniguchi, MD, Principal Investigator — Taniguchi Pediatrics Clinic; Hidehisa Shinohara, MD, Principal Investigator — Shinohara Pediatrics Clinic; Michiko Tanabe, MD, Principal Investigator — Tanabe Pediatrics Clinic; Haruo Kuroki, MD, Principal Investigator — Sotobo Children's Clinic; Hirokazu Sato, MD, Principal Investigator — Sunrise Children's Clinic; Katsumi Yamada, MD, Principal Investigator — Yamada Clinic; Hiroshi Sakiyama, MD, Principal Investigator — Sakiyama Pediatric Clinic; Hiroji Okawa, MD, Principal Investigator — Okawa Children & Family Clinic; Junichi Ito, MD, Principal Investigator — Ito ENT Clinic; Masato Morimoto, MD, Principal Investigator — MORIMOTO ENT CLINIC; Masakazu Umemoto, MD, Principal Investigator — Umemoto Pediatric Clinic; Tadashi Matuda, MD, Principal Investigator — Matsuda Pediatrics Clinic; Sadayoshi Torigoe, MD, Principal Investigator — Aquair Medical Station; Shigeru Mori, MD, Principal Investigator — Momotaro Clinic; Yutaka Fujimaki, MD, Principal Investigator — Fujimaki Ent Clinic; Masaki Kato, MD, Principal Investigator — Kato Ear Nose Throat Clinic; Hisakuni Sekino, MD, Principal Investigator — Sekino Hospital; Toshikazu Nagakura, MD, Principal Investigator — Yoga Allergy Clinic; Ichiro Ogiwara, MD, Principal Investigator — Ogiwara Ent Clinic; Akitoshi Funato, MD, Principal Investigator — Medical corporation Seisyuukai Funato Clinic; Naohisa Hoshino, MD, Principal Investigator — Medical corporation Ryoshukai Kanauchi Medical Clinic; Munechika Noguchi, MD, Principal Investigator — Social medical corporation IHL ShinagawaEastOne Medical Clinic; Chiaki Noguchi, MD, Principal Investigator — Shinkoiwa Ekimae Sougou Clinic; Kimihiko Yukisada, MD, Principal Investigator — Yukisada Clinic for internal disease; Hiroshi Shimomura, MD, Principal Investigator — Medical corporation Junyokai Musashino General Clinic; Mitsuhiro Nemoto, MD, Principal Investigator — Nemoto-geka-seikeigeka; Naoki Kawai, MD, Principal Investigator — Kawai Naika Iin; Shigehiro Yazima, MD, Principal Investigator — Yajima Children's Clinic; Tetsuhiko Nagao, MD, Principal Investigator — Midorino Clinic; Kenjiro Nakamura, MD, Principal Investigator — Tenjin Sogo Clinic; Wataru Ikematsu, MD, Principal Investigator — Kobori Building Clinic; Shiro Kimura, MD, Principal Investigator — Kimura Shiro Clinic; Mieko Ueda, MD, Principal Investigator — Ueda Naika Clinic; Minako Iwaya, MD, Principal Investigator — Iwaya Children's Clinic; Motohisa Ikeda, MD, Principal Investigator — Ikeda Naika Clinic; Tetsunari Maeda, MD, Principal Investigator — Sakura Clinic
Locations (38):
- Japan (38):
  - Research Site, Akashi-shi
  - Research Site, Chofu-shi
  - Research Site, Fuchu-shi
  - Research Site, Fujimi-shi
  - Research Site, Fukui-shi
  - Research Site, Fukuoka
  - Research Site, Fukuroi-shi
  - Research Site, Funabashi-shi
  - Research Site, Gifu
  - Research Site, Hatsukaichi-shi
  - Research Site, Hiroshima
  - Research Site, Ichikawa-shi
  - Research Site, Isumi
  - Research Site, Iwate-gun
  - Research Site, Katsushika-ku
  - Research Site, Kawasaki-shi
  - Research Site, Kisarazu-shi
  - Research Site, Kiyose-shi
  - Research Site, Kobe
  - Research Site, Koga-shi
  - Research Site, Kumamoto
  - Research Site, Kunitachi-shi
  - Research Site, Kuwana-shi
  - Research Site, Matsudo-shi
  - Research Site, Minatoku
  - Research Site, Morioka
  - Research Site, Nakano
  - Research Site, Okayama
  - Research Site, Ōta-ku
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Setagaya-ku
  - Research Site, Shinjuku-ku
  - Research Site, Shizuoka
  - Research Site, Taito-ku
  - Research Site, Toshima-ku
  - Research Site, Tsu
  - Research Site, Yokkaichi-shi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 1369 consented, 68 were excluded after screening.
Groups:
- MEDI3250: MEDI3250, 0.2mL as nasal spray
- Placebo: Placebo, 0.2mL as nasal spray
Period: Overall Study
Arm/Group | MEDI3250 | Placebo
Started | 868 | 433
Received IP (Safety Population) | 868 | 433
Per Protocol Population | 849 | 430
Completed | 865 | 432
Not Completed | 3 | 1
Not completed — Meet Exclusion Criteria No. 17 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MEDI3250 | Placebo | Total
Number analyzed (Participants) | 868 | 433 | 1301
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.0 (3.0) | 10.8 (2.8) | 10.9 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 408 | 226 | 634
  Male | 460 | 207 | 667
Number of Doses of Study Vaccine to be Received [Number; unit: Participants]
  1 | 841 | 421 | 1262
  2 | 27 | 12 | 39
Prior Influenza Vaccination [Number; unit: Participants]
  Yes | 788 | 386 | 1174
  No | 80 | 47 | 127

OUTCOME MEASURES:

1. Primary Outcome: the Incidence of Laboratory-confirmed Influenza Infection (Matched Strain)
Description: The vaccine efficacy of MEDI3250 compared to placebo against the incidence of laboratory-confirmed influenza infection (matched strain)
Time Frame: through the end of the influenza surveillance period, up to end Apr (6 months)
Population: Per Protocol Population
Measure: Number; unit: Participants
Arm/Group | MEDI3250 | Placebo
Number analyzed (Participants) | 849 | 430
Participants | 0 | 1
Statistical Analysis 1: Comparison: MEDI3250 vs Placebo; Test type: Superiority or Other; Exact conditional method — No statistical tests were used, instead the confidence interval was used for showing superiority. If lower bound of the 95% CI is greater than 0%, the efficacy of MEDI3250 is demonstrated; Estimated by an exact conditional method in total number of cases which follows a Poisson assumption; Vaccine efficacy (%) = 100.0, 95% CI 2-sided [-1875.3 to 100.0] — Vaccine efficacy (%) = (1-RR)*100 where RR = Risk Reduction

2. Secondary Outcome: the Incidence of Laboratory-confirmed Influenza Infection (Any Strain)
Description: The vaccine efficacy of MEDI3250 compared to placebo against the incidence of laboratory-confirmed influenza infection (any strain)
Time Frame: through the end of the influenza surveillance period, up to end Apr (6 months)
Measure: Number; unit: Participants
Arm/Group | MEDI3250 | Placebo
Number analyzed (Participants) | 849 | 430
Participants | 169 | 118
Statistical Analysis 1: Comparison: MEDI3250 vs Placebo; Test type: Superiority or Other; Exact conditional method — [p-value comment as in outcome 1, analysis 1]; Estimated by an exact conditional method in total number of cases which follows a Poisson assumption; Vaccine efficacy (%) = 27.5, 95% CI 2-sided [7.4 to 43.0] — Vaccine efficacy (%) = (1-RR)*100 where RR = Risk Reduction

3. Secondary Outcome: the Incidence of Laboratory-confirmed Influenza Infection (Matched Strain, by Strain)
Description: The vaccine efficacy of MEDI3250 compared to placebo against the incidence of laboratory-confirmed influenza infection (matched strain, by strain)
Time Frame: through the end of the influenza surveillance period, up to end Apr (6 months)
Population: Per Protocol Population
Measure: Number; unit: Participants
Arm/Group | MEDI3250 | Placebo
Number analyzed (Participants) | 849 | 430
Participants
  Strain A_H1N1 | 0 | 0
  Strain A_H3N2 | 0 | 0
  Strain B_Yamagata | 0 | 1
  Strain B_Victoria | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs experienced from administration of investigational product through 28 days post last vaccination were collected
Arm/Group | MEDI3250 | Placebo | Total Number
Serious Adverse Events (participants affected / at risk) | 3/868 | 3/433 | 6/1301
Other Adverse Events (participants affected / at risk) | 126/868 | 67/433 | 193/1301
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI3250 (N=868) | Placebo (N=433) | Total Number (N=1301)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.01% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI3250 (N=868) | Placebo (N=433) | Total Number (N=1301)
nasopharyngitis (Infections and infestations) | 70 (70) | 36 (36) | 106 (106)
rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 9 (9) | 23 (23)
upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 8 (8) | 26 (26)
Bronchitis (Infections and infestations) | 5 (5) | 7 (7) | 12 (12)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 2 (2) | 11 (11)
Diarrhoea (Gastrointestinal disorders) | 10 (10) | 5 (5) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less